CLINICAL TRIAL: NCT00000302
Title: Expanded Steady-State Pharmacokinetic Study, Comparing Liquid and Tablet Buprenorphine Formulations
Brief Title: Study Comparing Liquid and Tablet Buprenorphine Formulations - 5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-09260-5; P50-09260-5
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2005-11-07 (Estimated); Status verified 2002-12

CONDITIONS: Heroin Dependence
MeSH Terms: conditions — Heroin Dependence | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to compare liquid and tablet buprenorphine formulations.

DETAILED DESCRIPTION:
Participants were inducted on either liquid or tablet buprenorphine, in a double-blind, double-dummy manner. They each reached a steady state by the second week, and were scheduled to have blood draws in weeks 3, 4, 7, 8, 11, 12, 15, and 16.

ELIGIBILITY:
Inclusion Criteria:

M/F ages 21-50. Opiate dependence according to DSM-IV criteria. Currently enrolled in the outpatient protocol comparing liquid and tablet formulations of Buprenorphine. Agreeable to conditions of study and signed informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nursing women. Dependence on ETOH or benzodiazepines or other sedative-hypnotics. Acute hepatitis. Other medical conditions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0

PRIMARY OUTCOMES:
Drug use
Retention
Drug craving

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States